CLINICAL TRIAL: NCT04386824
Title: Comparison of Erectile Dysfunction and Optical Coherence Tomography Angiography Findings in Patients With Non Ocular Behçet's Disease
Brief Title: Erectile Dysfunction in Patients With Non Ocular Behçet's Disease
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Ayan, Assoc Prof, Dr, Antalya Training and Research Hospital
Other Study IDs: Descriptive
Record Dates: First submitted 2020-05-02; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Behçet Disease; Behcet Syndrome; Erectile Dysfunction
Keywords: Behçet's disease; erectile dysfunction
MeSH Terms: conditions — Behcet Syndrome; Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Behçet's disease: Male patients who arediagnosed as Behçet's disease according to International Study Group Classification Criteria
  Interventions: Other: Erectil dysfunction

INTERVENTIONS:
Other: Erectil dysfunction — A complete ophthalmological examination including best-corrected visual acuity using the decimal system (BCVA), measurement of intraocular pressure (IOP) and axial length (AL), slit-lamp examination and dilated fundus examination
  Other Names: Ophthalmological Examination

SUMMARY:
It was aimed to demonstrate whether erectile dysfunction is affected by BH pathogenesis and whether there is a relationship between erectile dysfunction and BD pathogenesis by assessing both sexual function and retinal micro-vascular blood flow in BH which may involve vessels from all calibrations and nature.

DETAILED DESCRIPTION:
Patients with factors and results that could cause sexual dysfunction will be excluded from the study.An International Index of ErectileFunction (IIEF) questionnaire will be applied to a total of 35 patients under 45 years old who met the inclusion criteria. IIEF's erectile function,sexual desire,sexual satisfaction,orgasmic function and general satisfaction sub parameters and Optical Coherence Eye Tomography (OCTA) data will compared.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of Behçet Disease
* No comorbid disease known to be associated with erectile dysfunction, including hypertension and diabetes mellitus
* Not overweight or obese (BMI≤25 kg/m2)
* Non-smokers
* No alcohol and/or substance abuse
* No known psychiatric disorder

Exclusion Criteria:

* prostatic disorder
* medication that may influence on erectile function (antihistamines, ß-blockers, etc.)
* sacroiliac joint or chronic articular involvement
* family history of glaucoma

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male with Behçet's patients
Study Population: Behçet's disease (BD) is a chronic, multi-systemic vasculitis characterized by remissions and exacerbations, where etiology hasn't been fully elucidated [1]. It was first described as oral aphthae, genital ulcerations, and iridocyclitis with hypopyon by Hulusi Behçet in 1937 [2]. Although its etiology hasn't been fully understood, it is widely accepted that the disease is caused by excessive inflammatory response triggered by environmental factors in individuals with genetic susceptibility
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function-15 | 1 week
  This scale assessing the quality of erectile function within the previous 4 weeks was developed by Rosen et al. in 1997. The Turkish validity study was performed by Turunç et al. [30]. The IIEF-15 assesses male sexual function in 5 domains: erectile function (1-30 points), orgasmic function (0-10 points), sexual desire (2-10 points), sexual satisfaction from intercourse (0-15 points) and overall satisfaction (2-10 points). In contrast to other functions, the severity of erectile dysfunction can be rated with an overall score ranging from 6 to 30 points. Erectile function was graded as follows: 0-10 points as severe erectile dysfunction (ED); 11-16 points as moderate ED; 17-21 points as mild-moderate ED; 22-25 points as mild ED; 26-30 points as no erectile dysfunction.
Optical coherence tomography angiography | 1 week
  It is a functional method that detects the movement contrast in the bloodstream and displays the capillary nets of the retina and choroid and the outer retina without using paint.It is a non-invasive method that provides static volumetric angiography information.From the quantitative measurement results presented by calculating automatically by the software used by the device, the area of the foveal avascular zone (PHASE), the value of the asymmetric index (AI), the superficial and Vascular density (VD) percentages and retinal thickness values in deep capillary plexuses were included in the study.OCTA findings are classified in stages 1-5. OCTA findings worsen as the stage number increases. While stage 1 shows normal superficial capillary plexus; In stage 5, decreased vascular density in the outer retina and significant thinning in the retina are observed.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ayan, Dr., Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Tarining and Research Hospital Ethics Commitee, Antalya, Muratpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Plan will be shared with Statistical Package for the Social Sciences version 20.

REFERENCES:
- [Result] Direskeneli H. Autoimmunity vs autoinflammation in Behcet's disease: do we oversimplify a complex disorder? Rheumatology (Oxford). 2006 Dec;45(12):1461-5. doi: 10.1093/rheumatology/kel329. Epub 2006 Sep 23. No abstract available. PMID 16998234